CLINICAL TRIAL: NCT02888197
Title: A Non-Interventional Extension Study to Investigate Vulvovaginal Candidiasis Recurrence and Candida Colonization Following a Phase 2 Randomized, Active-Controlled Study of Two Formulations of CD101 Compared to Fluconazole for the Treatment of Moderate to Severe Episodes of Acute Vulvovaginal Candidiasis
Brief Title: Non-Interventional Extension to Investigate Recurrence of Vulvovaginal Candidiasis and Candida Colonization
Status: Completed | Type: Observational
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CD101.TP.2.02
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Candidiasis, Vulvovaginal; Yeast Infection; Mycoses; Moniliasis, Vulvovaginal; Vaginitis, Monilial
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Candida isolates
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-interventional extension study to investigate VVC recurrence and candida colonization following the P2 acute VVC study

DETAILED DESCRIPTION:
Following completion of the Phase 2, multicenter, randomized, active-controlled study of the safety and tolerability of two formulations of CD101 compared to fluconazole for the treatment of moderate to severe episodes of acute vulvovaginal candidiasis (NCT07299432), subjects without a recurrence of VVC will be followed up to an additional 90 days +/- 14 days to assess candida colonization and recurrence of VVC.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in and completed the primary study through the Day 28 visit.
* Received at least one dose of study drug in the primary study
* Able to give written informed consent prior to completion of the primary study

Exclusion Criteria:

* Received systemic or topical vaginal non-study antifungal therapy at any time during the primary study
* Diagnosed with bacterial vaginosis, trichomonas, gonorrhea, chlamydia, or active herpes at any point during the primary study
* The Principal Investigator considers that the subject should not participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females previously enrolled in the primary study (NCT07299432) who had not been diagnosed with recurrence of vulvovaginal candidiasis and successfully completed the Day 28 visit in the primary study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Time to recurrence of clinical signs/symptoms of VVC | Up to Day 90 +/- 14 days
  Time to recurrence of clinical signs/symptoms of VVC

SECONDARY OUTCOMES:
Rate of candida colonization | Up to Day 90 +/- 14 days
  Rate of candida colonization
Rate of recurrence of clinical signs/symptoms of VVC | Up to Day 90 +/- 14 days
  Rate of recurrence of clinical signs/symptoms of VVC
Time to recurrence of culture confirmed VVC | Up to Day 90 +/- 14 days
  Time to recurrence of culture confirmed VVC
Rates of recurrence of culture confirmed VVC | Up to Day 90 +/- 14 days
  Rates of recurrence of culture confirmed VVC

CONTACTS AND LOCATIONS:
Overall Officials: Alena Jandourek, MD, Study Director — Cidara Therapeutics
Locations (23):
- United States (23):
  - Precision Trials AZ, Phoenix, Arizona
  - The Women's Clinical, P.A., Little Rock, Arkansas
  - Women's Health Care Research Corp, San Diego, California
  - Olympian Clinical Research, Clearwater, Florida
  - Women's Medical Research, Clearwater, Florida
  - Altus Research Inc, Lake Worth, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Augusta University, Augusta, Georgia
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Wayne State University, Detroit, Michigan
  - Saginaw Valley Medical Research Group LLC, Saginaw, Michigan
  - Lawrence OB GYN Clinical Research LLC, Lawrenceville, New Jersey
  - Alliance Women's Research Group LLC, Riverside Park, New Jersey
  - Soffolk OB/GYN, Port Jefferson, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Hawthorne Medical Research Inc, Winston-Salem, North Carolina
  - Unified Women's Clinical Research - Hickory, Winston-Salem, North Carolina
  - Women's Health Research, Columbus, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - TMC Life Research Inc., Houston, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Tidwewater Physicians for Women, Norfolk, Virginia
  - Seattle Women's Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided